CLINICAL TRIAL: NCT02598817
Title: Acceptability of "High Sn-2" Infant Formula in Non-Breast Fed Healthy Term Infants Regarding Gastrointestinal Tolerability by Both Parents and Pediatrician. An Open Label Pilot Study Evaluation in the Gulf Cooperation Council (GCC) Countries.
Brief Title: Acceptability and Gastrointestinal Tolerance of a High-Sn-2 Infant Formula
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 15.17.INF.ME
Record Dates: First submitted 2015-10-28; First posted 2015-11-06 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Infant Term Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard Infant Formula: Standard Infant Formula containing High Sn-2
  Interventions: Other: Standard Infant Formula

INTERVENTIONS:
Other: Standard Infant Formula — Standard Infant Formula containing High Sn-2

SUMMARY:
The purpose of this study is to evaluate the effects of term infant formula containing high 2-palmitic vegetable oil on stool composition, stool characteristics and gastrointestinal (GI) Tolerance.

DETAILED DESCRIPTION:
This is a multicenter, open label, observation study; 500 formula fed infants are planned to be enrolled from a network of general pediatricians in the Gulf countries (UAE, Kuwait, Qatar, and KSA). Eligible infants will consume a high sn-2 palmitate infant formula for 12 weeks. All enrolled infants will be evaluated at enrollment and at 4 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Formula fed healthy full term infants with normal birth weight (2500g 4000g)
* Partially breast and formula fed infants who drink at least 2 formula feedings per day; each to be at least 30ml
* Infants of both genders at age of 2 weeks to 12 weeks
* Infants of parents providing written informed consent before any study related activities are carried out

Exclusion Criteria:

* Preterm or IUGR babies
* Contraindication of standard infant formula
* Infants who have allergy of cow's milk protein
* Infants with Serious medical or surgical GI disease
* Infants with multiple congenital anomalies
* Infants with suspected chromosomal or metabolic disorder
* Infants of mothers with a health condition or socioeconomic problems that may interfere with their ability to take care of their infants
* Infants of parents who refuse to participate in the study

Ages: 2 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 500 healthy, full-term, formula fed infants
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Infant Stool Form Scale | 12 weeks
  frequency and consistency

SECONDARY OUTCOMES:
Changes from baseline to 12 weeks in Height centile | 12 weeks
  height (cm)
Changes from baseline to 12 weeks in Weight centile | 12 weeks
  weight(kg) and respective Wt z-scores
Changes from baseline to 12 weeks in Head Circumference centile | 12 weeks
  Head circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Islam Tawfiq Al Baroudi, MD, Principal Investigator — Pediatric Gastroenterologist
Locations (5):
- Saudi Arabia (3):
  - Tadawi General Hospital, Dammam
  - Almana Hospital, Jubail
  - Al Mouasat Hospital, Riyadh
- United Arab Emirates (2):
  - Sheikh Khalifa Medical City, Abu Dhabi
  - Al Garhoud Private Hospital, Dubai